CLINICAL TRIAL: NCT00310154
Title: ZD-1839 (Iressa®) With Concurrent Docetaxel and Conformal Three Dimensional Thoracic Radiation Followed by Consolidative Docetaxel and ZD-1839 for Patients With Stage III Non Small Cell Lung Cancer: A Phase I Study
Brief Title: Gefitinib, Docetaxel, and Radiation Therapy in Treating Patients With Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000466391; P30CA012197 (NIH); CCCWFU-62202; ZENECA-IRUSIRES0043; CCCWFU-BG03-310
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2011-11

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; large cell lung cancer; squamous cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma, Bronchiolo-Alveolar; Adenocarcinoma of Lung | interventions — Docetaxel; Gefitinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: docetaxel
Drug: gefitinib
Other: laboratory biomarker analysis
Radiation: radiation therapy

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving gefitinib together with docetaxel and radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of docetaxel when given together with gefitinib and radiation therapy in treating patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of docetaxel that can be safely delivered in combination with gefitinib and a definitive course of 3-D planned thoracic radiotherapy in patients with stage III non-small cell lung cancer.

OUTLINE: This is a dose-escalation study of docetaxel.

* Chemoradiotherapy: Patients receive concurrent chemoradiotherapy comprising docetaxel IV over 30 minutes on day 1 and thoracic radiotherapy once daily on days 1-5 in weeks 1-7 in the absence of disease progression or unacceptable toxicity.
* Consolidation chemotherapy: Beginning 2 weeks after the completion of chemoradiotherapy, patients receive consolidation chemotherapy comprising docetaxel IV over 60 minutes on days 1 and 22.
* Gefitinib therapy: Patients also receive oral gefitinib once daily beginning at the start of chemoradiotherapy and continuing for up to 1 year* in the absence of disease progression.

NOTE: *Patients continue to receive gefitinib during the 2-week rest period between chemoradiotherapy and consolidation chemotherapy.

Cohorts of 3-6 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Tumor tissue is tested to determine correlation between epidermal growth factor receptor presence and response to treatment.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 45 patients will be accrued in this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), including any of the following:

  * Squamous cell carcinoma
  * Adenocarcinoma (including bronchoalveolar cell)
  * Large cell anaplastic carcinoma (including giant and clear cell carcinomas)
* Stage IIIA/B disease

  * Unresectable disease
  * Tumors adjacent to a vertebral body allowed

    * No demonstrable bone invasion
    * All gross disease must be able to be encompassed in the radiation boost field in accordance with the homogeneity criteria
  * Contralateral mediastinal disease (N3) allowed if all gross disease can be encompassed in the radiation boost field in accordance with the homogeneity criteria

    * No scalene, supraclavicular, or contralateral hilar node involvement
  * Pleural effusion allowed if it is transudate, cytologically negative, and non-bloody AND tumor can be encompassed within a reasonable field of radiotherapy

    * No exudative, bloody, or cytologically malignant effusions
    * Pleural effusion seen on chest CT scan but not on chest x-ray and too small to tap allowed
* Measurable disease, defined as lesions that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan

  * No nonmeasurable disease, including any of the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
    * Tumor lesions situated in a previously irradiated area

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Granulocyte count ≥ 1,500/mm^3
* Hemoglobin > 8.0 g/dL
* Platelet count ≥ 100,000/mm^3
* Bilirubin < 1.5 mg/dL
* Creatinine < 1.5 times upper limit of normal (ULN)
* Meets 1 of the following criteria:

  * AST and ALT < 2 times ULN
  * AST and ALT ≤ 2.5 times ULN AND alkaline phosphatase (AP) normal
  * AST and ALT normal AND AP ≤ 4 times ULN
* FEV_1 ≥ 1.2 L
* No other currently active malignancy except nonmelanoma skin cancers

  * Patients are not considered to have another currently active malignancy if they have completed therapy for the other malignancy and are considered by their physician to be at < 30% risk of relapse (i.e., after treatment for early-stage prostate cancer)
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after completing treatment
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No known severe hypersensitivity to gefitinib or any of the excipients of this product
* No evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* No evidence of any other significant clinical disorder or laboratory finding that would limit compliance with study requirements
* No evidence of clinically active interstitial lung disease (asymptomatic, chronic stable radiographic changes allowed)
* No peripheral neuropathy ≥ grade 1

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior formal exploratory thoracotomy
* No prior chemotherapy or radiotherapy for NSCLC
* No prior epidermal growth factor-targeting drugs (i.e., gefitinib, erlotinib, or cetuximab)
* No other investigational agent within 30 days of study entry
* No concurrent phenytoin, carbamazepine, rifampicin, barbiturates, or Hypericum perforatum (St John's wort)
* No other concurrent hormonal therapy or chemotherapy except for the following:

  * Steroids for adrenal failure, allergic reactions, or septic shock
  * Hormones for nondisease-related conditions (e.g., insulin for diabetes)
  * Glucocorticosteroids as anti-emetics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2003-11; Primary Completion 2007-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To determine the feasability of daily ZD1839 delivered with concurrent 3-dimensional planned thoracic radiation | baseline to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Arthur William Blackstock, MD, Study Chair — Wake Forest University Health Sciences; Antonius A. Miller, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Center B, Petty WJ, Ayala D, Hinson WH, Lovato J, Capellari J, Oaks T, Miller AA, Blackstock AW. A phase I study of gefitinib with concurrent dose-escalated weekly docetaxel and conformal three-dimensional thoracic radiation followed by consolidative docetaxel and maintenance gefitinib for patients with stage III non-small cell lung cancer. J Thorac Oncol. 2010 Jan;5(1):69-74. doi: 10.1097/JTO.0b013e3181c59a0e. PMID 20035186